CLINICAL TRIAL: NCT02486354
Title: Safety and Efficacy of Icotinib in Advanced Metastatic Patients With NSCLC Previously Treated With Chemotherapy: a Single-arm, Phase 3 Study
Brief Title: Icotinib in Advanced Metastatic Patients With NSCLC Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-III01-V2
Record Dates: First submitted 2015-06-28; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- icotinib (Experimental): Patients were administered with oral icotinib (tablet form, 125 mg) three times daily within two days after enrollment until disease progression or unacceptable toxicity.
  Interventions: Drug: icotinib

INTERVENTIONS:
Drug: icotinib — Patients were administered with oral icotinib (tablet form, 125 mg) three times daily within two days after enrollment until disease progression or unacceptable toxicity.
  Other Names: Conmana

SUMMARY:
This study was a single-arm, multi-center, prospective, phase 3 trial aimed to evaluate the efficacy and safety of icotinib in patients with locally advanced or metastatic NSCLC after failure of at least one platinum-based chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced/metastatic (stage IIIB/stage IV, using the American Joint Committee on Cancer [AJCC] 6th edition of tumor-node-metastasis [TNM] staging system) NSCLC patients
* Progressed after at least one platinum-based chemotherapy regimen at entry
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* At least one measurable lesion by Response Evaluation Criteria in Solid Tumors version 1.0
* Adequate hematologic and biochemical values

Exclusion Criteria:

* Patients with symptomatic brain metastases
* Malignant tumor within the previous five years
* Severe infection; congestive heart failure
* Previous treatment with drugs targeting EGFR
* History of interstitial lung disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 6 months

SECONDARY OUTCOMES:
overall survival | 12 months
objective response rate | 2 months
number of patients suffered adverse events | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Study Chair — Cancer Hospital Chinese Academy of Medical Science
Locations (10):
- China (10):
  - Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Bejing Cancer Hospital, Beijing, Beijing Municipality
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Third Affiliated Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Sun yat-sen Univerisity Cancer Center, Guanzhou, Guangdong
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Result] Shi Y, Zhang L, Liu X, Zhou C, Zhang L, Zhang S, Wang D, Li Q, Qin S, Hu C, Zhang Y, Chen J, Cheng Y, Feng J, Zhang H, Song Y, Wu YL, Xu N, Zhou J, Luo R, Bai C, Jin Y, Liu W, Wei Z, Tan F, Wang Y, Ding L, Dai H, Jiao S, Wang J, Liang L, Zhang W, Sun Y. Icotinib versus gefitinib in previously treated advanced non-small-cell lung cancer (ICOGEN): a randomised, double-blind phase 3 non-inferiority trial. Lancet Oncol. 2013 Sep;14(10):953-61. doi: 10.1016/S1470-2045(13)70355-3. Epub 2013 Aug 13. PMID 23948351
- [Derived] Hu X, Zhang L, Shi Y, Zhou C, Liu X, Wang D, Song Y, Li Q, Feng J, Qin S, Xv N, Zhou J, Zhang L, Hu C, Zhang S, Luo R, Wang J, Tan F, Wang Y, Ding L, Sun Y. The Efficacy and Safety of Icotinib in Patients with Advanced Non-Small Cell Lung Cancer Previously Treated with Chemotherapy: A Single-Arm, Multi-Center, Prospective Study. PLoS One. 2015 Nov 24;10(11):e0142500. doi: 10.1371/journal.pone.0142500. eCollection 2015. PMID 26599904